CLINICAL TRIAL: NCT07406529
Title: Fostering Prosocial Behaviours Against Infectious Diseases Through Awe: A Randomized Controlled Trial
Brief Title: Fostering Prosocial Preventive Behaviours Through Awe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Qiuyan Liao, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Socialconhealth2025
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Infectious Diseases
Keywords: preventive behaviour; infectious diseases; awe
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be randomly assigned to study conditions using the automated randomization function of the online survey platform. Both participants and researchers will be blind to group allocation during data collection. Allocation information will only be revealed to the research team at the data analysis stage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention is a three-step mini game named Hidden Picture Puzzle (HPP) designed to induce the feeling of awe. In the game, participants will first see a picture of nature covered by six opaque blocks. They will be asked to guess the content of the picture. After making their choice, participants will be instructed to click the six blocks to gradually uncover the picture. Once all six blocks are removed, the full image will be revealed. In the final step, participants will be instructed to imagine themselves in the scene and describe their feelings by selecting the word from a provided list. To ensure that participants will have sufficient time to complete the imagination tasks, they will be required to pause for at least 15s before proceeding to indicate their immediate feeling. Each participant will complete four rounds of this mini game, each with a different picture.
  Interventions: Behavioral: Awe intervention
- Control group (Placebo Comparator): For the control group, the HPP will also follow a three-step format, identical in structure to the intervention condition. However, the images provided will depict everyday objects (e.g., a sofa or a bottle) rather than nature scenes. Similarly, when participants are asked to guess the content of the picture. After the participants finish uncovering the pictures, they will be asked to imagine their interaction with these daily objects and describe the features of the objects by selecting a word from a provided list. As in the intervention group, participants in the control group will complete four rounds of the mini game, each with a different image.
  Interventions: Behavioral: Neutral imagination

INTERVENTIONS:
Behavioral: Awe intervention — The intervention is a three-step mini game named Hidden Picture Puzzle (HPP) designed to induce the feeling of awe. In the game, participants will first see a picture of nature covered by six opaque blocks. They will be asked to guess the content of the picture. After making their choice, participants will be instructed to click the six blocks to gradually uncover the picture. Once all six blocks are removed, the full image will be revealed. In the final step, participants will be instructed to imagine themselves in the scene and describe their feelings by selecting the word from a provided list. To ensure that participants will have sufficient time to complete the imagination tasks, they will be required to pause for at least 15s before proceeding to indicate their immediate feeling. Each participant will complete four rounds of this mini game, each with a different picture.
  Arms: Intervention group
Behavioral: Neutral imagination — For the control group, the HPP will also follow a three-step format, identical in structure to the intervention condition. However, the images provided will depict everyday objects (e.g., a bottle) rather than nature scenes. Similarly, when participants are asked to guess the content of the picture. After the participants finish uncovering the pictures, they will be asked to imagine their interaction with these daily objects and describe the features of the objects by selecting a word from a provided list. As in the intervention group, participants in the control group will complete four rounds of the mini game, each with a different image.
  Arms: Control group

SUMMARY:
The goal of this randomized control trial is to investigate the impact pf awe on prosocial preventive behaviours against infectious diseases among adults from Hong Kong, Singapore, and ten major cities in Mainland China (Beijing, Shanghai, Guangzhou, Shenzhen, Hangzhou, Chongqing, Chengdu, Wuhan, Xi'an, Nanjing). The main questions it aims to answer are:

* Does experiencing awe increase adults' intentions to engage in prosocial preventive behaviours against infectious diseases, including vaccination, mask wearing, and social distancing?
* Does the impact vary across three research sites?

DETAILED DESCRIPTION:
This study will be conducted as a nested sub-study within a main longitudinal study implemented online. The baseline assessment of the longitudinal study was conducted between October and November 2025. Participants who agreed to be recontacted will be invited to join the randomized controlled trial (RCT) approximately four months after the baseline assessment, in February-March 2026. At that time, participants will be randomized in a 1:1 ratio into either the intervention or control group.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years) who live in
* Hong Kong, Singapore, and ten major cities in Mainland China (Beijing, Shanghai, Guangzhou, Shenzhen, Hangzhou, Chongqing, Chengdu, Wuhan, Xi'an, Nanjing) over the past one year
* Able to read and understand written Chinese or English
* Have access to the internet through computers, mobile phones, or tablets

Exclusion Criteria:

* Individuals with cognitive or linguistic difficulties that would prevent them from completing an online survey will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Intentions to participate in future preventive behaviours | Immediately after they complete the game with manipulation
  Participants will be asked their intentions to participate in future vaccination, mask wearing, and social distancing during next winter influenza season.
Behavioural choices in the pandemic vignettes | Immediately after they complete the game with manipulation
  Based on a hypothetical infectious disease pandemic, six vignettes will be shown to the participants, comprising three on vaccination and three on social distancing. Each vignette illustrates a trade-off between personal cost and social benefit in engaging in these prosocial behaviours. Participants will be asked to report how likely will they are to engage in the prosocial preventive behaviours.

SECONDARY OUTCOMES:
Intentions to engage in social activities | Immediately after they complete the game with manipulation
  Participants will also be asked their intentions to pengage in social activities.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong School of Public Health, Hong Kong, Hong Kong